CLINICAL TRIAL: NCT06217887
Title: Efficacy Comparison of Polyethylene Glycol Loxenatide and Gliclazide on the Brain Function in T2DM Patients: a Randomized, Parallel Controlled Clinical Trial
Brief Title: Efficacy Comparison of Polyethylene Glycol Loxenatide and Gliclazide on the Brain Function in T2DM Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Yan Bi, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: z-2017-26-1902
Record Dates: First submitted 2023-12-20; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes Mellitus; Cognitive Function Abnormal
Keywords: Functional MRI; Cognition; Olfactory function; loxenatide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognition Disorders | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- loxenatide Group (Experimental): loxenatide will be initiated and maintained at 0.2mg once weekly until the completion of the study. Meanwhile, all patients will also continue on their existing dose and regimen of metformin throughout the study. Visits at 4-week intervals will be performed to evaluate the safety of drugs. Metformin dose can be reduced in response to hypoglycaemia, but loxenatide could not be adjusted. If the plasma glucose still not achieve the target at the maximum dose, the maximum dose will be maintained until the completion of the study.
  Interventions: Drug: loxenatide Group
- Gliclazide Group (Experimental): Gliclazide will be initiated and maintained at 30mg/ day every morning until the completion of the study. Meanwhile, all patients will also continue on their existing dose and regimen of metformin throughout the study. Visits at 4-week intervals will be performed to evaluate the safety of drugs. Metformin dose can be reduced in response to hypoglycaemia, but Gliclazide could not be adjusted. If the plasma glucose still not achieve the target at the maximum dose, the maximum dose will be maintained until the completion of the study.
  Interventions: Drug: Gliclazide Group

INTERVENTIONS:
Drug: loxenatide Group — Loxenatide will be initiated and maintained at 0.2mg once weekly until the completion of the study. All patients will also continue on their existing dose and regimen of metformin throughout the study.
  Other Names: metformin
  Arms: loxenatide Group
Drug: Gliclazide Group — Gliclazide will be initiated and maintained at 30mg/day every morning. If necessary, the dose can be increased to 120mg once daily. All patients will also continue on their existing dose and regimen of metformin throughout the study.
  Other Names: metformin
  Arms: Gliclazide Group

SUMMARY:
This is a prospective, randomized, open label, parallel,4-month study to explore and evaluate the therapeutic effects of polyethylene glycol loxenatide on the cognitive function, olfactory function, and odor-induced brain activation in T2DM patients with normal cognitive status or MCI.

DETAILED DESCRIPTION:
This is a prospective, randomized, open label, parallel, 4-month study to explore and evaluate the therapeutic effects of polyethylene glycol loxenatide on the cognitive function, olfactory function, and odor-induced brain activation in T2DM patients with normal cognitive status or MCI inadequately controlled with metformin monotherapy. The control group was treated with Gliclazide. There are 1 principal investigator, 6 sub-investigators and 1 nurse in research centre. The sub-investigators will screen in the outpatient and inpatient departments to enroll 58 patients (29 patients for each arm) totally with the inclusion and exclusion criteria in 9 months. The patients will be randomized at a 1:1 ratio into loxenatide and Gliclazide treatment group with a computer-generated random order. All patients will also continue on their existing dose and regimen of metformin throughout the study. At the baseline, clinical information collection, 100g-steamed bread meal test, biochemical measurement, body composition analysis, cognitive assessment, olfactory test and functional magnetic resonance imaging(fMRI) scan will be conducted for all patients. During the treatment period, visits at 4-week intervals will be performed to evaluate the safety of drugs and adjust the dose of metformin if hypoglycaemia occurs; meanwhile, fasting and 2-hour postprandial plasma glucose assayed by fingerstick, physical examination, and olfactory test will be conducted. At the end of the study, all of the assessments will be performed again for all recruited subjects, including early withdrawal patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes mellitus ;
* Aged:40 -75 years ;
* Cognitive function assessment suggests normal status or mild cognitive impairment;
* a stable dose of metformin monotherapy (≥1,500 mg daily) for at least 90 days,
* HbA1c 7 - 10%;
* ≥6 years of education;
* Right-handed.

Exclusion Criteria:

* patients unable to complete brain MRI scanning;
* nasal disease that affected olfactory function;
* hepatic dysfunction with liver transaminases > 2.5 times upper normal limits and renal impairment with an estimated glomerular filtration rate < 60ml/min/1.73m2 ;
* acute cardio/cerebrovascular disease, psychiatric disorders, pancreatitis, acute infection, malignant tumor,thyroid disease and homorne drug use;
* a history of related drug allergy;
* alcohol or drug misuse;
* pregnant, breast-feeding or intending to become pregnant.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-05-10 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change of olfactory brain activation by fMRI | from baseline to 4-month follow-up
  Whether the activation degree of olfactory task fMRI brain area in the two groups after intervention was different from that before treatment and the difference of changes between the two groups. All patients underwent odor-induced task fMRI on a 3.0T MR scanner with 222 volumes for task fMRI and 230 volumes for resting-state fMRI. The odor-induced task consisted of "fresh air" "rest" and "scent". Odor-induced brain activation was assessed by a general linear model using Statistical Parametric Mapping 12 (SPM12) software. Following extraction of the three separate conditions "fresh air," "scent," and "rest" from the whole sequence, contrasts were made for each participant between "fresh air > rest" and "scent > rest." Odor-induced fMRI data were analyzed in the mask of the olfactory network, including the regions of bilateral parahippocampus, amygdala, piriform cortex, insula, orbitofrontal cortex, hippocampus, and entorhinal cortices.

SECONDARY OUTCOMES:
Change of cognitive function | from baseline to 4-month follow-up
  Cognitive function were improved, which means MoCA scores were improved after treatment, the RBANS total score increased by 0.5 standard deviation compared with baseline after treatment.
Change of metabolism | from baseline to 4-month follow-up
  The changes of glycosylated hemoglobin among the two groups before and after intervention. The level of glycosylated hemoglobin <7% means better glucose metabolism.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Zhang Z, Zhang B, Wang X, Zhang X, Yang QX, Qing Z, Zhang W, Zhu D, Bi Y. Olfactory Dysfunction Mediates Adiposity in Cognitive Impairment of Type 2 Diabetes: Insights From Clinical and Functional Neuroimaging Studies. Diabetes Care. 2019 Jul;42(7):1274-1283. doi: 10.2337/dc18-2584. Epub 2019 May 21. PMID 31221697
- [Background] Cheng H, Zhang Z, Zhang B, Zhang W, Wang J, Ni W, Miao Y, Liu J, Bi Y. Enhancement of Impaired Olfactory Neural Activation and Cognitive Capacity by Liraglutide, but Not Dapagliflozin or Acarbose, in Patients With Type 2 Diabetes: A 16-Week Randomized Parallel Comparative Study. Diabetes Care. 2022 May 1;45(5):1201-1210. doi: 10.2337/dc21-2064. PMID 35263425